CLINICAL TRIAL: NCT00121797
Title: Risk Factors for Postpartum Bacteruria, Does Labor Cause UTI?
Brief Title: Peripartum Bacteruria and Urinary Tract Infections (UTI)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 26-5.9.03-HMO-CTIL; Women's health grant 8060101
Record Dates: First submitted 2005-07-17; First posted 2005-07-21 (Estimated); Last update posted 2006-11-07 (Estimated); Status verified 2005-07

CONDITIONS: Urinary Tract Infection
Keywords: Postpartum Period
MeSH Terms: conditions — Urinary Tract Infections

INTERVENTIONS:
Procedure: urine culture
Drug: antibiotics according to culture

SUMMARY:
In the last years urinary tract infections (UTI) and pyelonephritis have been the most common reason for readmission to our hospital after birth. UTI is know to be one of the leading causes of postpartum fever affecting about 3%-8% of all postpartum women.

The investigators hypothesize that collecting urine cultures pre- and postnatally may help identify women at risk for developing UTI, while treating women with positive cultures could decrease the rehospitalization rate due to postpartum fever. Collecting data during delivery may help identify women at risk for this complication.

DETAILED DESCRIPTION:
The study is planned as a randomized controlled study with 500 women in each arm. The study group will have pre and post labor urine cultures taken, and the risk factors during delivery will be documented, while the control group will have no cultures taken, as the common practice prior to the study.

Women with positive cultures will be contacted by telephone, and antibiotic treatment recommended according to bacteria sensitivity. All women will be contacted by telephone 1 month post partum and data regarding urinary tract symptoms and need for hospitalization, will be collected. The rehospitalization rate will be documented and compared between the two groups.

The assumption is that routine urine culture to women in the peripartum period may reduce the UTI rate and hospitalization after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Parturients planned for vaginal delivery

Exclusion Criteria:

* Parturients receiving antibiotic treatment during delivery or in the week before

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2004-01; Study Completion 2005-06 (Estimated)

PRIMARY OUTCOMES:
Rate of rehospitalization for postpartum fever
Incidence of UTI in the early puerperium

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Elram, MD, Principal Investigator — Hadassah Medical Organization
Locations (2):
- Israel (2):
  - Clinical microbiology, Hadassah Ein-Kerem Medical centre, Jerusalem
  - Obs&Gyn Hadassah Ein-Kerem Medical center, Jerusalem